CLINICAL TRIAL: NCT03457051
Title: A Randomized Trial Comparing Outcomes of Unicompartmental and Total Knee Replacement for Isolated Medial Osteoarthritis: A Feasibility Study
Brief Title: Unicompartmental Knee Arthroplasty (UKA) Versus Total Knee Arthroplasty (TKA) of Medial Osteoarthritis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of study funding
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OHREB # 20120904-01H
Record Dates: First submitted 2014-11-28; First posted 2018-03-07 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Knee Arthroplasty (TKA) (Active Comparator): In total (complete) knee arthroplasty (TKA), the orthopaedic surgeon removes the damaged areas of the knee and replaces the components with an artificial joint that is made of plastic or metal.
  Interventions: Procedure: Total Knee Arthroplasty (TKA)
- Unicompartmental Knee Arthroplasty (UKA) (Experimental): Unicompartment (partial) knee arthroplasty (UKA) has been available for over 40 years and differs from TKA in that only the most affected and symptomatic compartment (most commonly medial, but occasionally lateral and patella femoral) are replaced
  Interventions: Procedure: Unicompartmental Knee Arthroplasty (UKA)

INTERVENTIONS:
Procedure: Total Knee Arthroplasty (TKA) — In total (complete) knee arthroplasty (TKA), the orthopaedic surgeon removes the damaged areas of the knee and replaces the components with an artificial joint. The device that will be used is: Stryker TKA Triathlon system implant Cruciate retaining radius femur design. This device has been approved for use by Health Canada.
  Arms: Total Knee Arthroplasty (TKA)
Procedure: Unicompartmental Knee Arthroplasty (UKA) — Unicompartment (partial) knee arthroplasty (UKA) has been available for over 40 years and differs from TKA in that only the most affected and symptomatic compartment (most commonly medial, but occasionally lateral and patella femoral) are replaced. The device that will be used is: Stryker PKR implant cemented and fixed bearing design. This device has been approved for use by Health Canada.
  Arms: Unicompartmental Knee Arthroplasty (UKA)

SUMMARY:
This study allows patients to take part of the decision making between a unicompartment knee (partial ) or a total Knee replacement . Using the measures of a decision aid questionnaire which explicitly details the risks and benefits of both procedures.The study will use subjective (reported by patient) and objective data (which will be measured) to allow the determination if one option is superior to the other. Information gathered from this study will be used to assist future patients in selecting the surgical option that best fits their life style.

A feasibility pilot study of a randomized clinical trial will help to evaluate the outcomes of both procedures and help shape a multicentre Canadian study.

DETAILED DESCRIPTION:
Osteoarthritis of the knee is an increasingly common problem for many Canadians aged 50 or greater. When conservative management fails, patients are often offered a type of knee replacement as treatment. The choices are a total knee replacement or a partial knee replacement, which carry distinct advantages and disadvantages. Typically, patients with partial knee replacement have less post operative pain, quicker recovery and enhanced function with greater knee bend. There is however a higher chance of revision where the pain is not relieved or the implant fails. The decision for which replacement to offer is now primarily surgeon driven, shaped by their experience, review of evidence and capability to perform either of these options. Canadian patients would benefit from a decision making model so their own values can shape and determine the decision. This research hopes to evaluate the merits of a patient based decision aid which explicitly details the risks and benefits of both procedures as they are best understood today. Further, the quality of the current evidence is only moderately strong limited by patient selection biases and there is a need for contemporary comparative study trial of the 2 procedures to help clinicians and patients make the decision.

A feasibility pilot study of a randomized clinical trial is being proposed to evaluate the outcomes of both procedures, which will help shape a multicentre Canadian study.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria must and will be restricted to those patients who are generally considered candidates for UKA. Specific inclusion criteria will be restricted to patients:

* Who report that most of their pain (greater than 75%) is located in the medial part of the knee on a regular basis.
* With active range of motion from 10° of extension to 100° of flexion.
* With an intact, competent, anterior cruciate ligament.
* With overall limb alignment correctable to neutral, indicating a competent medial collateral ligament.
* With radiographs showing primarily bone-on-bone disease in the medial compartment with minimal wear in both the lateral and patellofemoral compartments of the knee.
* 50 to 80 years of age.
* With a Body Mass Index (BMI) less than 40.

For the secondary outcome of motion analysis, only patients exhibiting the following characteristics will be suitable for assessment:

* BMI of 35 or less
* No other ipsilateral or contralateral lower limb joint disorders

Exclusion Criteria:

* Those with inflammatory arthritis
* Those with no fixed address
* Those unable to commit to study requirements and follow-ups

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index | 36 months
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire is the sum of WOMAC A (total pain), WOMAC B (stiffness) and WOMAC C (functional impairment) subscores. All the items are scored on a scale of 0-4; lower scores are indicative of lower disease burden. Values are summed for a combined WOMAC score (Total score ranges from 0-96, with higher scores indicating worse pain, stiffness, and functional limitations).

SECONDARY OUTCOMES:
Change in Oxford Knee Score (OKS) | 36 months
  Patient-reported questionnaire. The sum of the questionnaire will be totaled. Oxford Knee Score Scale range 0 (severe arthritis) - 48 (satisfactory joint function)
Change in Knee Society Score (KSS) | 36 months
  The Knee Society Score (KSS) is comprised of 4 components: 1) An "Objective" Knee Score (7 items: 100 points), 2) A Patient Satisfaction Score (5 items: 40 points), 3) A Patient Expectation Score (3 items: 15 points), and 4) A Functional Activity Score (19 items: 100 points). Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Quantitative analysis of gait using EMG and motion capture | 12 months
  A ten-camera infrared motion capture system will be used to track patients gait in a Biomechanics Laboratory. Retroreflective markers will be placed on the body in various locations to track muscle activity. Patients will be asked to perform 5 trials of level walking, 5 trials of inclined and declined walking (12.5% slope), 5 trials of going up and down stairs and 5 trials of sitting and standing motions. Only patients exhibiting the following characteristics will be suitable for assessment: BMI of 35 or less, No other ipsilateral or contralateral lower limb joint disorders.
Short Term Recovery | 6 months
  Patients recovery will be evaluated using the 40 item, quality of recovery (QoR-40) questionnaire. The sum of all scores (the total) will be reported (Minimum=40, Maximum=200). Higher scores are indicative of better perceived recovery while lower scores are associated with a worse perceived recovery.
Clinical Measures | 6months
  Patient complications (if any) will be recorded by the surgeon during post-operative clinical assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Dervin, MD,MSc,FRCSC, Principal Investigator — OHRI / The Ottawa Hospital/ University of Ottawa
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No